CLINICAL TRIAL: NCT04759417
Title: A Multi-center Prospective Observational Study to Evaluate and Compare Diagnostic Accuracy and Reliability of Variables of the CHOKAI and STONE Scores to Predict the Presence of Ureteric Stones as Confirmed on CT Scans
Brief Title: Comparison of CHOKAI vs STONE Score to Predict the Presence of Ureteric Stones in Patients With Renal Colic: A Multi-center Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: Zayed Military Hospital (Other Government)
Responsible Party: Principal Investigator, Mohammad Anzal Rehman, Emergency Medicine Resident, Zayed Military Hospital
Other Study IDs: SEHA-019
Record Dates: First submitted 2021-02-03; First posted 2021-02-18 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Ureteric Stone
Keywords: ureteric stone; CHOKAI; STONE; UAE; renal colic
MeSH Terms: conditions — Ureterolithiasis; Renal Colic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: The STONE score has traditionally been used as a clinical prediction tool to predict the presence of ureteric stones in patients presenting with renal colic. More recently, the CHOKAI score was introduced and found to have superior diagnostic accuracy on both internal and external validation.

Objective: Our study aims to externally validate and compare the use of both the CHOKAI and STONE score in a population of UAE patients presenting to the Emergency Department for renal colic.

Methods: Over a period of approximately 6 months, the study will follow Emergency Department Physicians at each institution and retrieve data from their encounters with patients presenting with renal colic. Parameters for both CHOKAI and STONE scores will be logged, extracted and matched against a reference standard of CT scan to compare diagnostic accuracy of both scores to predict the presence of ureteric stones in this population.

Goals: Evaluation of the findings will discern applicability of scores to the UAE population and contribute to reducing unnecessary radiation exposure.

To our knowledge, no studies have compared the use of these scores to diagnose urolithiasis in the United Arab Emirates. Furthermore, this will be the first study to externally validate the CHOKAI score outside of Japan using a controlled, prospective design.

DETAILED DESCRIPTION:
Over a period of approximately 6 months, the study will follow Emergency Department Physicians at each of three separate institutions and retrieve data from their encounters with patients presenting with renal colic. Parameters for both CHOKAI and STONE scores will be logged, extracted and matched against a reference standard of CT scan to compare diagnostic accuracy of both scores to predict the presence of ureteric stones in this population

Full-time ED Physicians from each institution will be recruited to participate in the study as follows:

Each ED Physician shall be provided with Data Collection Sheet. This form will provide them with a standardized option to enter the components of the STONE and CHOKAI score using data normally conducted in the history taking and physical examination of patients suspected to have ureteric stones. Additional items have also been included to investigate for other variables that could influence clinical prediction of presence of ureteric stones.

Those patients suspected to have ureteric stones will have confirmation of urolithiasis by non-contrast CT scan. Though the investigators will log the data in their respective data collection sheets per patient, they will not be involved in entering this data onto the study's database.

Data will be collected for a period of approximately 6 months from February 1, 2021 onward, with a target sample size of 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult population (≥18 years of age) presenting to the Emergency Department with symptoms determined by the investigating ED Physician to be suspicious of urolithiasis (e.g. flank pain, lower abdominal pain, back pain and/or hematuria)
* Patients suspected to have ureteric stone who underwent CT scan to confirm diagnosis

Exclusion Criteria:

Complicated ureteric colic:

* Abnormal vital signs - body temperature > 37.7 °C or systolic blood pressure ˂90 mmHg)
* Active malignancy
* Abnormal kidney function (abnormal levels of creatinine/BUN)
* Recent (within past 6 months) trauma or urologic surgery
* Age <18 years
* Pregnant patient
* Patient with incomplete interview/documentation data (e.g. missing US/CT/ UA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the Emergency Department with symptoms suspicious of urolithiasis
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy comparison | 6 months
  Compare the diagnostic accuracies of the CHOKAI and STONE scores in predicting the presence of ureteric stones by using differences in the area under the curve (AUC) between the CHOKAI and STONE scores, calculated using Receiver Operating Characteristic (ROC) analysis

SECONDARY OUTCOMES:
Determine optimal cut-off point | 6 months
  Point on ROC analysis where maximum sensitivity and specificity exist. Calculate sensitivity, specificity, positive likelihood ratio and negative likelihood ratio at this point
Rate of admission for patients | 6 months
  Frequency of admission disposition for patients, to evaluate for any association of high risk on predictor scores to admission dispositions

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Anzal Rehman, MD, Principal Investigator — Zayed Military Hospital
Locations (3):
- United Arab Emirates (3):
  - Sheikh Shakhbout Medical City, Abu Dhabi
  - Tawam Hospital, Abu Dhabi
  - Zayed Military Hospital, Abu Dhabi

IPD SHARING:
Plan to Share IPD: Yes
The protocol for selection of patients used for prospective data collection shall be made available for the entirety of the study duration, including the Informed Consent Form we will use during patient encounters. The Statistical Analysis Plan (SAP) will be shared after results are compiled (approximately in 6 months from study start date) and processed by the biostatistician for a period of 3 months
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol and Informed Consent data will be available for 6 months from study start date Study Analysis Plan (SAP) will be available for 3 months once data collection is completed and results compiled for analysis
Access Criteria: Any interested researcher can approach the Principal Investigator, Mohammad Anzal Rehman, at chokai.study@outlook.com for any of the details listed above within the time frames mentioned for access to the same.